CLINICAL TRIAL: NCT03258814
Title: Treat and Train - A Post-Marketing-Observational Study (PMOS) to Determine the Effectiveness of Combined Adalimumab Treatment and Active Supervised Training in Patients With Axial Spondyloarthritis
Brief Title: A Post-Marketing-Observational Study (PMOS) to Determine the Effectiveness of Combined Adalimumab Treatment and Active Supervised Training in Patients With Axial Spondyloarthritis (axSpA)
Acronym: Treat & Train
Status: Terminated | Type: Observational
Why Stopped: Low or No Enrollment
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-710
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-08

CONDITIONS: Axial Spondyloarthritis
Keywords: axial spondyloarthritis; active supervised training; physical training; adalimumab; spinal mobility; physiotherapy; physical function; health-related quality of life; pain; disease activity; psychosocial risk factors; workability; Bath Ankylosing Spondylitis Metrology Index (BASMI)
MeSH Terms: conditions — Axial Spondyloarthritis; Pain | interventions — Standard of Care; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active Supervised Training (AST): Participants with axSpA and treated with adalimumab (HUMIRA®) according to the local product label and local standard of care were to receive active supervised and standardized training (AST).
  Interventions: Behavioral: Active Supervised Training (AST)
- Standard of Care (SOC) Physiotherapy: Participants with axSpA and treated with adalimumab (HUMIRA®) according to the local product label and local standard of care were to receive standard of care physiotherapy, according to the physiotherapist discretion.
  Interventions: Behavioral: Standard of Care (SOC) Physiotherapy

INTERVENTIONS:
Behavioral: Active Supervised Training (AST) — The active supervised and standardized training consisted of 24 units of exercise within 20 weeks performed in certified training centers and was focused on back fitness, core strengthening and patient engagement to treat back pain and functional impairment.
  Groups: Active Supervised Training (AST)
Behavioral: Standard of Care (SOC) Physiotherapy — Standard of care physiotherapy as used in this study included active as well as passive training and massages according to the physiotherapist discretion.
  Groups: Standard of Care (SOC) Physiotherapy

SUMMARY:
This study is a non-interventional, longitudinal and non-confirmatory study to compare an active supervised training (AST) with standard of care (SOC) physiotherapy in patients with axial spondyloarthritis and stable response to adalimumab (HUMIRA®) with respect to health-related outcomes. The primary objective is the improvement in spinal mobility after a 6 month training program.

DETAILED DESCRIPTION:
Treatment of axSpA patients with adalimumab (HUMIRA®) was according to the local adalimumab product label and local standard of care. AxSpA patients who responded to newly initialized adalimumab treatment based on physicians' decision, and who were eligible for active physiotherapy were enrolled in the study. Although this was a non-interventional study, participants were randomly assigned to receive either active supervised and standardized training physiotherapy or standard of care physiotherapy in order to provide adequate numbers of participants in each comparison group.

Participants who consented to participate in the study were observed for up to 12 months from Baseline (defined as the Randomization visit where participants were assigned to one of the two physiotherapy options).

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with axial spondyloarthritis (axSpA) (either ankylosing spondylitis (AS) or non-radiographic axial spondyloarthritis (nr-axSpA)), fulfilling the Assessment of Spondyloarthritis International Society (ASAS) classification, aged at least 18 years
* Prescription of Humira® (adalimumab) for treating axSpA according to the local product label
* Eligibility for active physiotherapy according to the rheumatologist and physiotherapist
* Participants must have signed written informed consent before starting any study related assessments or procedures.

Exclusion Criteria:

* Participants with total spinal ankylosis based on the investigators' assessments of available radiographs
* Participants who are not eligible for active supervised training or active physiotherapy at the discretion of the rheumatologist and/or the physiotherapist
* Participants with poorly controlled medical condition(s), which in the opinion of the investigator, would put the participant at risk by participation in the protocol
* Any prior treatment with a biologic disease-modifying antirheumatic drugs (DMARD) is prohibited.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with axial spondyloarthritis who received Humira® per local product label at rheumatology centers in Germany.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (6):
- Germany (6):
  - Rheumahaus Studien GbR, Potsdam, DE /ID# 164494, Potsdam, Brandenburg
  - MVZ Wittenbergplatz PP Orthos /ID# 204802, Berlin
  - Rheumapraxis /ID# 164461, Halle
  - Praxis Ortho DE /ID# 204149, Hamburg
  - Praxis internistische Rheumato /ID# 164463, Leipzig
  - Krankenhaus St. Josef /ID# 164501, Wuppertal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with axial spondyloarthritis (AS) at 7 study sites in Germany. Eligible participants were receiving treatment with adalimumab (HUMIRA®) based on therapist's decision and local label requirements, must have had a response to adalimumab and have been eligible for active physiotherapy.
Pre-assignment Details: An enrollment period of treatment initiation and response assessment for 3 to 5 months preceded Randomization. This study was terminated early due to slow enrollment. Up to study termination 17 patients met all inclusion and none of the exclusion criteria and were enrolled in the study. A total of 7 of these patients were randomized into the study.
Groups:
- Active Supervised Training (AST): Participants were to receive active supervised and standardized training (AST).
- Standard of Care (SOC) Physiotherapy: Participants were to receive standard of care physiotherapy, according to the physiotherapist discretion.
- Not Randomized: Participants who were enrolled in the study but were not randomized.
Period: Overall Study
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy | Not Randomized
Started | 4 | 3 | 10
Completed | 0 | 0 | 0
Not Completed | 4 | 3 | 10
Not completed — Early Termination | 4 | 3 | 10

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 52 [37 to 66] | 31 [30 to 43] | 38 [30 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Bath Ankylosing Spondylitis Metrology Index (BASMI) [Mean (Standard Deviation); unit: units on a scale] — BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. The total score ranges from 0 to 10, reflecting mild to moderate disease activity and functional ability in the spinal column. The higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 2 | 2 | 4
    (all) | 2.9 (3.3) | 2.2 (0.8) | 2.6 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Change Form Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Month 6
Description: BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. The total BASMI score ranges from 0 to 10 reflecting mild to moderate disease activity and functional ability in the spinal column. The higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis
Time Frame: Baseline and Month 6
Population: No participants had a Month 6 visit due to early study termination, hence the primary endpoint could not be assessed.
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change Form Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Month 3
Description: as for outcome 1
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | 1.1 (0.4) |

3. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities, each on a numeric rating scale (NRS) ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher score indicating more limitations.
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -0.1 (0.1) |

4. Secondary Outcome: Change From Baseline in Assessment of Spondyloarthritis International Society (ASAS) Health Index (HI)
Description: The ASAS HI measures functioning and health across 17 aspects of health in patients with AS, including pain, emotional functions, sleep, sexual function, mobility, self care, and community life. The ASAS HI consists of 17 questions, each answered by the participant as agree (1) or disagree (0). The responses to the 17 dichotomous items are summed up to give a total score ranging from 0 to 17, with a lower score indicating a better and a higher score indicating an inferior health status.
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | 0.5 (0.7) |

5. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10 where lower scores indicate less disease activity.
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -0.4 (0.2) |

6. Secondary Outcome: Percentage of Participants Achieving a BASDAI 50 Response
Description: The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from baseline in BASDAI score.
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

7. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (C-reactive protein [CRP]) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity."
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -0.3 (0.1) |

8. Secondary Outcome: Percentage of Participants With ASDAS Inactive Disease
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity." The percentage of participants with ASDAS inactive disease, defined as ASDAS < 1.3, is reported.
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 50.0 |

9. Secondary Outcome: Percentage of Participants With ASDAS Low Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity." The percentage of participants with ASDAS low disease activity, defined as ASDAS < 2.1, is reported.
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 50.0 |

10. Secondary Outcome: Percentage of Participants With ASDAS Moderate Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity." The percentage of participants with ASDAS moderate disease activity, defined as an ASDAS ≥ 1.3 to < 2.1, is reported.
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

11. Secondary Outcome: Percentage of Participants With ASDAS High Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity." The percentage of participants with high disease activity, defined as an ASDAS ≥ 2.1 to < 3.5, is reported.
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 50.0 |

12. Secondary Outcome: Percentage of Participants With ASDAS Very High Disease Activity
Description: ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity." The percentage of participants with very high disease activity, defined as an ASDAS ≥ 3.5, is reported.
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

13. Secondary Outcome: Percentage of Participants Achieving ASDAS Major Improvement
Description: ASDAS Major Improvement is defined as a change from Baseline ≥ 2.0. ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity."
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

14. Secondary Outcome: Percentage of Participants Achieving ASDAS Clinically Important Improvement
Description: ASDAS clinically important improvement is defined as a change from Baseline ≥ 1.1.
  ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP) as an objective measure of inflammation. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS are: < 1.3 for "inactive disease"; ≥ 1.3 to < 2.1 for "moderate disease activity"; ≥ 2.1 to ≤ 3.5 for "high disease activity" and ≥ 3.5 for "very high disease activity."
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

15. Secondary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 20 Response
Description: ASAS20 response was defined as improvement of ≥ 20% relative to Baseline and absolute improvement of ≥ 1 unit (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 unit) in the potential remaining domain:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

16. Secondary Outcome: Percentage of Participants Achieving an ASAS 40 Response
Description: ASAS40 response was defined as improvement of ≥ 40% relative to baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration in the potential remaining domain:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

17. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission
Description: ASAS partial remission is defined as an absolute score of ≤ 2 units on a 0 to 10 scale for each of the four following domains:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (none) to 10 (severe);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Month 3
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
percentage of participants | 0.0 |

18. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Pain
Description: The patient's global assessment of pain was assessed on a NRS from 0 (no pain) to 10 (pain as bad as it could be).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -0.5 (0.7) |

19. Secondary Outcome: Change From Baseline in Patient's Assessment of Total Back Pain
Description: The patient's assessment of total back pain was assessed on a NRS from 0 (no pain) to 10 (most severe pain).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | 0.5 (0.7) |

20. Secondary Outcome: Change From Baseline in Patient's Assessment of Nocturnal Back Pain
Description: The patient's assessment of nocturnal back pain was assessed on a NRS from 0 (no pain) to 10 (most severe pain).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -0.5 (0.7) |

21. Secondary Outcome: Change From Baseline in Modified Work Ability Index (WAI)
Description: This is used to assess participant's work ability.
Time Frame: Baseline and Month 3
Population: No participants had available WAI data
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in Fatigue
Description: Fatigue was assessed as Question 1 of the BASDAI, on a NRS from 0 (none) to 10 (very severe).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -0.5 (0.7) |

23. Secondary Outcome: Change From Baseline in Severity and Duration of Morning Stiffness
Description: Morning stiffness was measured as the mean of the 2 morning stiffness-related BASDAI NRS scores:
  Question 5: Level of morning stiffness assessed by the patient on a scale from 0 (none) to 10 (very severe), and Question 6: Duration of morning stiffness assessed by the patient on a scale from 0 (0 hours) to 10 (2 hours or more duration).
Time Frame: Baseline and Month 3
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 2 | 0
scores on a scale | -1.5 (0.7) |

24. Secondary Outcome: Change From Baseline in Fear-Avoidance Belief Questionnaire Score (FABQ)
Description: The FABQ measures patients' fear of pain and consequent avoidance of physical activity because of their fear. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale, where 0 = completely disagree, 6 = completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Time Frame: Baseline and Month 3
Population: No participants had available FABQ data
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Active Supervised Training (AST) | Standard of Care (SOC) Physiotherapy | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 2/4 | 2/3 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Supervised Training (AST) (N=4) | Standard of Care (SOC) Physiotherapy (N=3) | Not Randomized (N=10)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early termination of the study, no interpretations or conclusions can be made based on the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT03258814/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03258814/SAP_001.pdf